CLINICAL TRIAL: NCT02507102
Title: A Feasibility Study of the Nativis Voyager® System in Patients With Recurrent Glioblastoma Multiforme (GBM) in Australia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nativis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAT-105
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigational Voyager Therapy (Experimental): Investigational treatment with Voyager Therapy
  Interventions: Device: Voyager

INTERVENTIONS:
Device: Voyager — Non-invasive RFE therapy

SUMMARY:
This feasibility study will assess the effects of the Nativis Voyager therapy in patients with recurrent GBM who have either failed standard of care or are intolerant to therapy. The study will enroll and treat up to eleven subjects over six months. Safety and clinical utility will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has histologically confirmed diagnosis of GBM.
2. Subject has failed or intolerant to radiotherapy.
3. Subjects has failed or intolerant to temozolomide therapy.
4. Subject has progressive disease with at least one measureable lesion on MRI or CT.
5. Subject is at least 18 years of age.
6. Subject has a KPS ≥ 60.
7. Subject has adequate organ and marrow function.
8. Subject has provided signed informed consent.

Exclusion Criteria:

1. Subject has life expectancy less than eight weeks
2. Subject has received other investigational therapy within the last 28 days.
3. Subject has received surgery within the last two weeks or not fully from prior surgery.
4. Subject has a clinically significant electrolyte abnormality.
5. Subject has an active implantable (e.g., neurostimulator, pacemaker) or other electromagnetic device.
6. Subject has a metal implant, including a stent, in the head or neck that is incompatible with MRI.
7. Subject is known to be HIV positive.
8. Subject is pregnant, nursing or intends to become pregnant during the study period.
9. Subject is participating in other investigational research.
10. Subject has any condition that at the discretion of the investigator would preclude participation in the study.
11. Subject is unable or unwilling to comply with the protocol-required follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Incidence and evaluation of any serious adverse events associated with the Nativis Voyager System | 6 months
Tumor Response | 2 months
  Tumor imaging response (RANO) at two months of therapy.

SECONDARY OUTCOMES:
Overall survival at six months compared with historical response | 6 months
Progression free survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Donna Morgan Murray, PhD, Study Director — Nativis, Inc.
Locations (1):
- St. Vincent's Hospital Melbourne, Melbourne, Victoria, Australia